CLINICAL TRIAL: NCT01497665
Title: A Phase II, Multi-center, Open-label Study Evaluating the Efficacy and Safety of GRN1005 in Non-Small Cell Lung Cancer Patients With Brain Metastases
Brief Title: GRN1005 in Non-Small Cell Lung Cancer (NSCLC) Patients With Brain Metastases (GRABM-L)
Acronym: GRABM-L
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Angiochem Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP1005B017
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC) With Brain Metastases
Keywords: GRN1005; ANG1005; LRP-1; Targeted Therapy; Brain Tumor; Blood Brain Barrier; Peptide-Drug Conjugate (PDC); Brain Metastases; Paclitaxel; Taxol; NSCLC; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — paclitaxel-Angiopep-2 conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GRN1005 alone (Experimental): GRN1005 alone
  Interventions: Drug: GRN1005

INTERVENTIONS:
Drug: GRN1005 — 650 mg/m2 IV every 3 weeks
  Other Names: ANG1005

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of GRN1005 in patients with brain metastases from non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult patients (≥ 18 years)
2. Histologically or cytologically-documented NSCLC (EGFR mutation status must be known)
3. Brain metastases from NSCLC, which:

   have radiologically-progressed after WBRT or are present without prior WBRT
4. At least one radiologically-confirmed and measurable lesion (≥ 1.0 cm in the longest diameter) within14 days prior to the first dose of GRN1005 (Cycle 1, Day 1), as follows: an intra-cranial disease lesion (≥ 1.0 cm in the longest diameter) confirmed by Gd-MRI, or an extra-cranial disease lesion (≥ 1.0 cm in the longest diameter) confirmed by MRI or CT scan with contrast Prior stereotactic radiosurgery (SRS) is allowed; however, metastatic brain lesions previously treated with SRS are not allowed as target or as non-target lesions.
5. Patients must be neurologically stable, defined as being on stable doses of corticosteroids and anticonvulsants (not EIAEDs, including phenytoin, phenobarbitol, carbamazepine, fosphenytoin, primidone, oxcarbazepine) for ≥ 5 days prior to obtaining the baseline Gd-MRI of the brain and ≥ 5 days prior to first dose of GRN1005 (Cycle 1, Day 1).
6. Karnofsky Performance Score (KPS) ≥ 80%
7. Completed WBRT for intra-cranial lesions ≥ 28 days prior to first dose of GRN1005 (with the exception of local radiation therapy for palliation to extra-cranial sites, i.e., bone). All clinically significant toxicities must have resolved to ≤ NCI CTCAE v4.0 Grade 1.0.

Key Exclusion Criteria:

1. NCI CTCAE v4.0 Grade ≥ 2 neuropathy
2. CNS disease requiring immediate neurosurgical intervention (e.g., resection, shunt placement, etc.)
3. Known intra-cranial hemorrhage
4. Known leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Lawrence, Study Director — Angiochem Inc; Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (9):
  - Univ. of California San Diego, La Jolla, California
  - Univ. Coloardo at Denver, Aurora, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern Univ., Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Univ. of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
- McGill Univ., Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GRN1005 Alone
Started | 16
Completed Effifcacy Assessment | 10 (Number of patients who completed efficacy assessment with CNS lesions per Overall RECIST 1.1.)
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1. Safety population (all patients): 16
  2. Efficacy population (defined as the number of patients who had ≥1 intracranial lesions followed as target or non-target lesions, and who were evaluated by Overall RECIST v.1.1):10
Arm/Group | GRN1005 Alone
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall (Intra-cranial and Extra-cranial) Objective Response Rate in Non-small Cell Lung Cancer (NSCLC) Patients With Brain Metastasis
Description: Tumor response was assessed by Gd-MRI for intracranial lesions and CT/MRI with contrast of chest, abdomen, pelvis for extracranial lesions using modified OVERALL RECIST v1.1 as follows: Complete Response (CR), disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions and non-target lesions stable or decreased; Stable Disease (SD), < 30% decrease but <20% increase in target lesions and non-target lesions stable or decreased; Progressive disease (PD), >= 20% (>= 5 mm) increase in the sum of diameters of the target lesions, taking as reference the smallest sum on study, non-target lesions increased or appearance of a new lesion; Overall Response (OR) = CR + PR.
Time Frame: upon enrollment through end of study period (1 year after last patient is enrolled)
Measure: Number; unit: participants
Arm/Group | GRN1005 Alone
Number analyzed (Participants) | 10
participants
  PR | 2
  SD | 3
  PD | 5

2. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Time Frame: Upon enrollment through end of study period (1 year after last patient is enrolled)
Measure: Number; unit: participants
Arm/Group | GRN1005 Alone
Number analyzed (Participants) | 16
participants | 16

3. Secondary Outcome: Duration of Overall Objective Response
Time Frame: Upon enrollment through end of study period (1 year after last patient is enrolled)
Population: Once the study was terminated, no further data on response was collected and there was insufficient number of participants with data collected for this outcome measure.
Arm/Group | GRN1005 Alone
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Overall Progression Free Survival
Time Frame: Upon enrollment through end of study period (1 year after last patient is enrolled)
Population: Once the study was terminated, no further efficacy data was collected and there was insufficient number of participants with data collected for this outcome measure.
Arm/Group | GRN1005 Alone
Number analyzed (Participants) | 0

5. Secondary Outcome: Six Month Overall Survival
Time Frame: Upon enrollment through end of study period (1 year after last patient is enrolled)
Population: Once the study was terminated, no further survival data was collected and there was insufficient number of participants with data collected for this outcome measure.
Arm/Group | GRN1005 Alone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: After informed consent, prior to initiation of GRN1005: only SAEs caused by a protocol-mandated intervention. After initiation of GRN1005: all AEs and SAEs until 30 days following the last administration of study drug.
Description: All SAEs and all Other (not including serious) AEs are reported regardless of attribution.
Arm/Group | GRN1005 Alone
Serious Adverse Events (participants affected / at risk) | 9/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GRN1005 Alone (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Mucosal inflammation (General disorders) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GRN1005 Alone (N=16)
Anemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 7
Thombocytopenia (Blood and lymphatic system disorders) | 3
Deafness (Ear and labyrinth disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Oedema peripheral (General disorders) | 4
Face edema (General disorders) | 2
Fatigue (General disorders) | 6
Mucosal inflammation (General disorders) | 4
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Hemorrhage intracranial (Nervous system disorders) | 1
Hypoesthesia (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 3
Dysphoria (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Nocturia (Renal and urinary disorders) | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 2
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Mucosal infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
White blood cell count increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Ataxia (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No